CLINICAL TRIAL: NCT06955078
Title: Effects of Visual Motor Integration on Visual Perception, Spatial Awareness and Motor Skills in Preschool Children
Brief Title: Effects of VMI on Visual Perception, Spatial Awareness and Motor Skills in Preschool Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/Hadeeqa Jabeen
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Preschool Children
Keywords: visual motor integration; preschool; visual perception; Beery-Buktenica Developmental Test of VMI

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trial performed in which 60 children equally divided into two groups and randomly allocated. Inclusion criteria for the study will be Children age 4 to 6 years old and all will be right-handed dominant with no history of visual or neurological abnormalities and exclusion criteria will be Children who presented a disability indicating a central nervous system dysfunction children age below 4 Years and above 6 years. One experimental group will perform Visual Motor Tasks, the other controlled group will perform routine class tasks. Pre and post assessment will be done. Outcomes to be analyzed will be enhancement in visual perception, spatial awareness and motor skills in preschool children by after performing VMI tasks. Data collection will be done before and after the intervention
Who Masked: Participant
Masking Description: Participants will get separate VMI training and possible efforts will be put to mask the both group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Visual motor integration Group): (Experimental): Group A will perform all the class along with the VMI tasks include:
  * Drawing (pictures and shapes for geometry)
  * Handwriting components-letter formation, sizing, spacing, and line orientation
  * Gross motor and PE activities the VP task will be used to measure an individual's visual abilities.
  * Discriminating and understanding left from right
  * Recognizing letters and numbers
  * Learning to read/write
  * Providing or obtaining directions
  * Visualizing objects or past experiences
  Visual skills can also impact a student's performance in the school setting as seen in the following:
  * Trouble discriminating left from right
  * Reversal of letter, numbers, or words when copying or writing
  * Mistaking words with similar beginnings when reading
  Interventions: Other: Visual Motor Integration
- Group B (No Intervention): Only class work will be done by the students.

INTERVENTIONS:
Other: Visual Motor Integration — The Beery Visual Motor Integration will be used to measure the integration of visual perception and motor skills as the participant children imitated and copied a developmentally sequential series of geometric forms using pencil and paper. As the task progressed, the levels of difficulty in geometric forms increased.
  VP task will be used to measure an individual's visual abilities without the integration of fine motor skills. Children will be asked to point to the item in the array, which was identical to the target figure. The choices will be written on answer sheets by experimenters or children themselves. Elapsed time will be recorded beginning with Item 7, and the task discontinued after 3 minutes. Children will be told to connect dots and to draw within provided borders. Elapsed time was recorded beginning with Item 7 and the task ended up after 5 minutes.
  Arms: Group A (Visual motor integration Group):

SUMMARY:
The preschool stage is an important period for children to develop their motor, language, cognitive, and social-emotional skills. pre-school years are the best time to intervene and correct developmental delays. VMI is linked to learning-related tasks like writing, measuring it in youngsters is essential. Earlier studies reported that children with deficits in VMI had lower academic achievements, the inadequate spatial organization of written work, and lower performance in mathematics and reading performance. The Beery-Buktenica Developmental Test of Visual-Motor Integration, Sixth Edition (Beery VMI-6), determined participants' VMI, VP and motor skills during the pre- and post-tests. Exposure to VMI tasks including, visual perception, spatial awareness and motor skills can be enhanced. VP is assessed by Visual Perception Task (VP Task) and Motor Coordination Task (MC Task) and spatial awareness is assessed by BAS 3.The aim of study is to analyze effects of VMI on visual perception, spatial awareness and motor skills in preschool children.

The current study will be randomized control trial; data will be collected from The Leaders Lyseum School Lahore. The study will include 60 children equally divided into two groups and randomly allocated. Inclusion criteria for the study will be Children age 4 to 6 years old and all will be right-handed dominant with no history of visual or neurological abnormalities and exclusion criteria will be Children who presented a disability indicating a central nervous system dysfunction children age below 4 Years and above 6 years. One experimental group will perform Visual Motor Tasks, the other controlled group will perform routine class tasks. Pre and post assessment will be done. Outcomes to be analyzed will be enhancement in visual perception, spatial awareness and motor skills in preschool children by after performing VMI tasks. Data collection will be done before and after the intervention. Tools used for data collection will be. Data will be analyzed through SPSS version 23.00.

DETAILED DESCRIPTION:
Group A Experimental (Visual motor integration Group): Group A will perform all the class along with the VMI tasks include:

* Drawing (pictures and shapes for geometry)
* Handwriting components-letter formation, sizing, spacing, and line orientation
* Writing fluency (speed and accuracy)
* Reproducing drawings, letters, etc. from the board or a book
* Understanding left and right or other directional concepts
* Gross motor and PE activities Visual Perception Task (VP Task) the VP task will be used to measure an individual's visual abilities.
* Discriminating and understanding left from right
* Matching objects or images
* Recognizing letters and numbers
* Providing or obtaining directions
* Visualizing objects or past experiences
* Developing eye-hand coordination

Group B Control group (Free play group): In this group only class work will be done no VMI tasks are assigned and performed. The participants will be assessed by using The Beery Visual Motor Integration 6th Edition will be used to measure the integration of visual perception and motor skills and VP task will be used to measure an individual's visual abilities.

ELIGIBILITY:
Inclusion Criteria:

* Children were 4 to 6 years old
* No history of visual or neurological abnormalities

Exclusion Criteria:

* • Children who presented a disability indicating a central nervous system dysfunction

  * Children wearing glasses

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-07-16 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) | 12 weeks
  Visual Motor Integration Task (VMI Task) The Beery VMI 6th Edition (33) will be used to measure the integration of visual perception and motor skills as the participant children imitated and copied a developmentally sequential series of geometric forms using pencil and paper. As the task progressed, the levels of difficulty in geometric forms increased.
  VP task will be used to measure an individual's visual abilities without the integration of fine motor skills. Children will be asked to point to the item in the array, which was identical to the target figure. The choices will be written on answer sheets by experimenters or children themselves.
Test of Spatial Assembly (TOSA) | 12 Weeks
  For each of the 2-D and 3-D portions of the TOSA, participants will receive a training trial followed by six test trials. During each test trial, the child will be shown a target figure composed of either 2-D geometric shapes or 3-D interlocking blocks. The child will be provided individual pieces, matching those in the target, and will be instructed to make their pieces look just like the target figure. The task required participants to exercise spatial visualization, shape decomposition and composition, and manual construction of complex shape forms in planar space and 3-dimensional space.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amjad, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin LY. Differences between preschool children using tablets and non-tablets in visual perception and fine motor skills. Hong Kong J Occup Ther. 2019 Dec;32(2):118-126. doi: 10.1177/1569186119888698. Epub 2019 Dec 6. PMID 32009863
- [Background] Bolger LE, Bolger LA, O'Neill C, Coughlan E, O'Brien W, Lacey S, Burns C, Bardid F. Global levels of fundamental motor skills in children: A systematic review. J Sports Sci. 2021 Apr;39(7):717-753. doi: 10.1080/02640414.2020.1841405. Epub 2020 Dec 30. PMID 33377417
- [Background] Prochaska E, Ammenwerth E. A Digital Box and Block Test for Hand Dexterity Measurement: Instrument Validation Study. JMIR Rehabil Assist Technol. 2023 Sep 15;10:e50474. doi: 10.2196/50474. PMID 37713251
- [Background] Oberer N, Gashaj V, Roebers CM. Motor skills in kindergarten: Internal structure, cognitive correlates and relationships to background variables. Hum Mov Sci. 2017 Apr;52:170-180. doi: 10.1016/j.humov.2017.02.002. PMID 28222343
- [Background] Flores P, Coelho E, Mourao-Carvalhal I, Forte P. Relationships between Math Skills, Motor Skills, Physical Activity, and Obesity in Typically Developing Preschool Children. Behav Sci (Basel). 2023 Dec 7;13(12):1000. doi: 10.3390/bs13121000. PMID 38131856
- [Background] Lopes L, Santos R, Pereira B, Lopes VP. Associations between gross motor coordination and academic achievement in elementary school children. Hum Mov Sci. 2013 Feb;32(1):9-20. doi: 10.1016/j.humov.2012.05.005. Epub 2012 Dec 20. PMID 23260614